CLINICAL TRIAL: NCT04129944
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Single-Dose Study of UBX0101 in Moderate to Severe, Painful Osteoarthritis of the Knee
Brief Title: A Study to Assess the Safety and Efficacy of a Single Dose of UBX0101 in Patients With Osteoarthritis of the Knee
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Unity Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UBX0101-MUS-201
Record Dates: First submitted 2019-10-15; First posted 2019-10-17 (Actual); Results first posted 2021-12-29 (Actual); Last update posted 2021-12-29 (Actual); Status verified 2021-11

CONDITIONS: Osteoarthritis, Knee
Keywords: Osteoarthritis; Painful Osteoarthritis; Osteoarthritis, Knee; Senescence
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo
- UBX0101 0.5 mg (Experimental)
  Interventions: Drug: UBX0101
- UBX0101 2.0 mg (Experimental)
  Interventions: Drug: UBX0101
- UBX0101 4.0 mg (Experimental)
  Interventions: Drug: UBX0101

INTERVENTIONS:
Drug: UBX0101 — Investigational drug intra-articular injection
  Arms: UBX0101 0.5 mg; UBX0101 2.0 mg; UBX0101 4.0 mg
Other: Placebo — Placebo intra-articular injection
  Arms: Placebo

SUMMARY:
A study to assess efficacy, safety, and tolerability of a single-dose intra-articular administration of UBX0101 in patients with moderate to severe painful knee osteoarthritis (OA).

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, single-dose, parallel-group study to assess the efficacy, safety, and tolerability of a single-dose intra-articular (IA) administration of UBX0101 in patients with moderate to severe painful knee osteoarthritis (OA).

Approximately 180 patients will be randomized (1:1:1:1) to one of four treatment groups (three dose levels of UBX0101 and Placebo; approximately 45 patients per group), all administered by IA route at Week 0. The four treatment groups will be enrolled concurrently.

The primary objective of the study is to evaluate the effect of IA administration of UBX0101 on the change from baseline to Week 12 of pain in the target knee.

ELIGIBILITY:
Key Inclusion Criteria:

* Patients who are ambulatory with a diagnosis of OA of the knee and who have baseline pain with a mean of ≥ 4 and ≤ 9 on the 11-point (0-10) average daily pain NRS for at least five of seven days during the Screening period.
* Kellgren-Lawrence grade of 1-4 on a weight-bearing radiograph of target knee.
* Patients aged ≥ 40 and ≤ 85 years.
* Patients are permitted but not required to use an oral NSAID, serotonin and norepinephrine reuptake inhibitors (SNRIs), tramadol, or acetaminophen, provided that they have been taking a stable dose and regimen of medication for at least 4 weeks prior to Screening.

Key Exclusion Criteria:

* Patients with any condition, including laboratory or imaging findings and findings in the medical history or in the pre-study assessments, that in the opinion of the Investigator or the Medical Monitor constitutes a risk or contraindication for participation in the study or that could interfere with the study objectives, conduct, or evaluation or prevent the patient from fully participating in all aspects of the study.
* Patients with a body mass index (BMI) ≥40 kg/m2 or a body habitus that precludes the MRI.
* Patients with fibromyalgia
* Systemic autoimmune disease with musculoskeletal involvement or any history of a systemic inflammatory arthritis
* Patients who have received IA treatment in the target knee with steroids or hyaluronic acid derivatives within the last 16 weeks prior to Screening, or with extended-release corticosteroid (e.g., Zilretta®) within the last 20 weeks
* Patients who are using a topical NSAID or topical analgesics on the target knee.
* Patients who have used opioid analgesics (other than tramadol), marijuana or marijuana-derived products (e.g., cannabidiol), and topical capsaicin on the target knee within 8 weeks prior to Screening
* Patients with a history of traumatic knee injury to the target knee, including, but not limited to, patients with meniscal root tear, within 2 years of study entry.
* Patients who have undergone diagnostic arthroscopy to the target knee in the previous 6 months.
* Patients who have undergone arthroscopic surgery (including microfracture and meniscectomy) on the target knee in the last 2 years prior to the Screening visit or are anticipated to have arthroscopic surgery on either knee at any time during the study period.
* Patients with a history of previous total or partial knee arthroplasty.
* Patients with an effusion at the Screening visit, which, in the opinion of the Investigator following examination and discussions with the patient, requires drainage for symptom relief.
* Patients who have had regenerative joint procedures on any joint, including, but not limited to, platelet-rich plasma injections, stem cell transplantation, autologous chondrocyte transplantation, or mosaicplasty.
* Patients with secondary arthritis that involves the target knee or would confound assessments of knee OA

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2019-10-30 (Actual); Primary Completion 2020-05-20 (Actual); Study Completion 2020-08-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — UNITY Biotechnology
Locations (20):
- United States (20):
  - Central Research Associates, Birmingham, Alabama
  - Coastal Clinical Research, LLC., Mobile, Alabama
  - Fiel Family and Sports Medicine, Tempe, Arizona
  - Tucson Orthopaedic Institute, Tucson, Arizona
  - Biosolutions Clinical Research Center, La Mesa, California
  - Diablo Clinical Research, Walnut Creek, California
  - Charter Research, Lady Lake, Florida
  - Well-Pharma Medical Research, Miami, Florida
  - Precision Clinical Research, Sunrise, Florida
  - Premier Medical Associates, The Villages, Florida
  - Chicago Clinical Research Institute, Chicago, Illinois
  - The Alliance for Multispecialty Research, Wichita, Kansas
  - Alliance for Multispecialty Research-Lexington, Lexington, Kentucky
  - The Alliance for Multispecialty Research, Kansas City, Missouri
  - Hassman Research Institute, Berlin, New Jersey
  - Albuquerque Clinical Trials, Albuquerque, New Mexico
  - Drug Trials America, Hartsdale, New York
  - Rochester Clinical Research, Rochester, New York
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Coastal Carolina Research Center, North Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | UBX0101 0.5 mg | UBX0101 2.0 mg | UBX0101 4.0 mg
Started | 46 | 45 | 46 | 46
Completed | 44 | 45 | 45 | 43
Not Completed | 2 | 0 | 1 | 3
Not completed — Death | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | UBX0101 0.5 mg | UBX0101 2.0 mg | UBX0101 4.0 mg | Total
Number analyzed (Participants) | 46 | 45 | 46 | 46 | 183
Age, Continuous [Median (Full Range); unit: years] | 65.0 [43.0 to 79.0] | 63.0 [43.0 to 80.0] | 66.0 [40.0 to 74.0] | 63.0 [42.0 to 81.0] | 64.0 [40.0 to 81.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 20 | 15 | 16 | 66
  Male | 31 | 25 | 31 | 30 | 117
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 5 | 9 | 3 | 28
  Not Hispanic or Latino | 35 | 40 | 37 | 43 | 155
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 8 | 11 | 8 | 11 | 38
  White | 38 | 34 | 37 | 34 | 143
  More than one race | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 12 of the Western Ontario and McMaster Universities Osteoarthritis Index Pain Subscale (WOMAC-A) Score in Patients Receiving a Single Dose of UBX0101 Versus Those Receiving Placebo
Description: WOMAC-A is assessed by a Likert scale on a range from 0 (none) to 4 (extreme), with higher scores indicating higher levels of pain
Time Frame: Baseline to Week 12
Population: Missing data for some subjects.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | UBX0101 0.5 mg | UBX0101 2.0 mg | UBX0101 4.0 mg
Number analyzed (Participants) | 46 | 45 | 46 | 46
score on a scale
  Baseline | 2.20 (0.577) | 2.05 (0.509) | 2.08 (0.658) | 2.11 (0.647)
  Week 12: number analyzed (Participants) | 43 | 45 | 46 | 43
  Week 12 | 1.12 (0.848) | 1.16 (0.731) | 1.04 (0.718) | 1.10 (0.707)
  Change in Score from Baseline to Week 12: number analyzed (Participants) | 43 | 45 | 46 | 43
  Change in Score from Baseline to Week 12 | -1.07 (0.924) | -0.89 (0.678) | -1.03 (0.884) | -1.03 (0.747)

2. Secondary Outcome: Change From Baseline to Week 12 of the Western Ontario and McMaster Universities Osteoarthritis Index Function Subscale (WOMAC-C) Score in Patients Receiving a Single Dose of UBX0101 Versus Those Receiving Placebo
Description: WOMAC-C is assessed by a Likert scale on a range from 0 (none) to 4 (extreme), with higher scores indicating higher levels of physical disability
Time Frame: Baseline to Week 12
Population: Missing data for some subjects.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | UBX0101 0.5 mg | UBX0101 2.0 mg | UBX0101 4.0 mg
Number analyzed (Participants) | 46 | 45 | 46 | 46
score on a scale
  Baseline | 2.26 (0.546) | 2.17 (0.527) | 2.16 (0.541) | 2.22 (0.660)
  Week 12: number analyzed (Participants) | 43 | 45 | 46 | 43
  Week 12 | 1.18 (0.812) | 1.11 (0.771) | 1.17 (0.772) | 1.24 (0.827)
  Change in Score from Baseline to Week 12: number analyzed (Participants) | 43 | 45 | 46 | 43
  Change in Score from Baseline to Week 12 | -1.07 (0.892) | -1.06 (0.770) | -0.99 (0.878) | -1.00 (0.772)

3. Secondary Outcome: Change From Baseline to Week 12 of the Weekly Mean of the Average Daily Pain (ADP) Intensity Scores on the 11-point Numeric Rating Scale (NRS) in Patients Receiving a Single Dose of UBX0101 Versus Those Receiving Placebo
Description: ADP is assessed by NRS on a range from 0 (no pain) to 10 (worst pain imaginable), with higher scores indicating higher levels of pain
Time Frame: Baseline to Week 12
Population: Missing data for some subjects.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | UBX0101 0.5 mg | UBX0101 2.0 mg | UBX0101 4.0 mg
Number analyzed (Participants) | 46 | 45 | 46 | 46
Score on a scale
  Baseline | 6.66 (1.382) | 6.48 (1.167) | 6.56 (1.463) | 6.68 (1.542)
  Week 12: number analyzed (Participants) | 41 | 40 | 42 | 38
  Week 12 | 3.48 (2.597) | 3.51 (2.262) | 3.67 (2.217) | 3.95 (2.029)
  Change in Score from Baseline to Week 12: number analyzed (Participants) | 41 | 40 | 42 | 38
  Change in Score from Baseline to Week 12 | -3.14 (2.626) | -3.05 (2.155) | -2.83 (2.452) | -2.63 (2.041)

4. Secondary Outcome: Change From Baseline (Over the Entire 24-week Period, Including Both the Primary Study Period and the 12-week Follow-up Period) to Week 24 for the WOMAC-A, NRS, and WOMAC-C Scores in Patients Receiving a Dose of UBX0101 Versus Those Receiving Placebo
Description: WOMAC-A is assessed by a Likert scale on a range from 0 (none) to 4 (extreme), with higher scores indicating higher levels of pain WOMAC-C is assessed by a Likert scale on a range from 0 (none) to 4 (extreme), with higher scores indicating higher levels of physical disability.
  Average Daily Pain (ADP) is assessed by Numerical Rating Score (NRS) on a range from 0 (no pain) to 10 (worst pain imaginable), with higher scores indicating higher levels of pain.
Time Frame: Baseline to Week 24
Population: Missing data for some subjects.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | UBX0101 0.5 mg | UBX0101 2.0 mg | UBX0101 4.0 mg
Number analyzed (Participants) | 46 | 45 | 46 | 46
score on a scale
  WOMAC-A Baseline | 2.20 (0.577) | 2.05 (0.509) | 2.08 (0.658) | 2.11 (0.647)
  WOMAC-A Week 24: number analyzed (Participants) | 44 | 45 | 45 | 43
  WOMAC-A Week 24 | 1.06 (0.872) | 1.04 (0.777) | 1.09 (0.683) | 1.12 (0.821)
  Change in WOMAC-A Score from Baseline to Week 24: number analyzed (Participants) | 44 | 45 | 45 | 43
  Change in WOMAC-A Score from Baseline to Week 24 | -1.12 (0.936) | -1.02 (0.711) | -1.00 (0.735) | -1.00 (0.884)
  WOMAC-C Baseline | 2.26 (0.546) | 2.17 (0.527) | 2.16 (0.541) | 2.22 (0.660)
  WOMAC-C Week 24: number analyzed (Participants) | 44 | 45 | 45 | 43
  WOMAC-C Week 24 | 1.14 (0.853) | 1.03 (0.803) | 1.17 (0.714) | 1.22 (0.848)
  Change in WOMAC-C Score from Baseline to Week 24: number analyzed (Participants) | 44 | 45 | 45 | 43
  Change in WOMAC-C Score from Baseline to Week 24 | -1.11 (0.902) | -1.13 (0.822) | -1.01 (0.736) | -1.00 (0.728)
  NRS Baseline | 6.66 (1.382) | 6.48 (1.167) | 6.56 (1.463) | 6.68 (1.542)
  NRS Week 24: number analyzed (Participants) | 24 | 29 | 32 | 27
  NRS Week 24 | 3.60 (2.317) | 3.14 (2.094) | 3.50 (2.171) | 3.52 (2.029)
  Change in NRS Score from Baseline to Week 24: number analyzed (Participants) | 24 | 29 | 32 | 27
  Change in NRS Score from Baseline to Week 24 | -3.01 (2.235) | -3.26 (2.139) | -3.22 (2.458) | -2.91 (2.412)

5. Secondary Outcome: Incidence of Treatment Emergent Adverse Events (TEAEs)
Time Frame: Baseline to Week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | UBX0101 0.5 mg | UBX0101 2.0 mg | UBX0101 4.0 mg
Number analyzed (Participants) | 46 | 45 | 46 | 46
Participants | 18 | 20 | 24 | 21

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Placebo | UBX0101 0.5 mg | UBX0101 2.0 mg | UBX0101 4.0 mg
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/45 | 0/46 | 1/46
Serious Adverse Events (participants affected / at risk) | 1/46 | 2/45 | 1/46 | 3/46
Other Adverse Events (participants affected / at risk) | 18/46 | 20/45 | 26/46 | 22/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=46) | UBX0101 0.5 mg (N=45) | UBX0101 2.0 mg (N=46) | UBX0101 4.0 mg (N=46)
Cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 1
Coronary Artery Disease (Cardiac disorders) | 0 | 0 | 0 | 1
Goitre (Endocrine disorders) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Knee arthroplasty (Surgical and medical procedures) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=46) | UBX0101 0.5 mg (N=45) | UBX0101 2.0 mg (N=46) | UBX0101 4.0 mg (N=46)
Atrial Fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0
Coronary Artery Disease (Cardiac disorders) | 0 | 0 | 0 | 1
Stress Cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Goitre (Endocrine disorders) | 0 | 1 | 0 | 0
Macular Degeneration (Eye disorders) | 0 | 0 | 1 | 0
Retinal Vein Occlusion (Eye disorders) | 0 | 0 | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Chest Discomfort (General disorders) | 0 | 0 | 2 | 0
Chest Pain (General disorders) | 0 | 1 | 0 | 0
Discomfort (General disorders) | 0 | 1 | 0 | 0
Injection Site Erythema (General disorders) | 1 | 0 | 0 | 0
Injection Site Irritation (General disorders) | 0 | 1 | 0 | 0
Injection Site Pruritus (General disorders) | 1 | 0 | 0 | 0
Oedema Peripheral (General disorders) | 0 | 1 | 0 | 0
Pain (General disorders) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0
Seasonal Allergy (Immune system disorders) | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 1 | 0
Chronic Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0
Covid-19 (Infections and infestations) | 0 | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 1 | 0
Ear Infection (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis Viral (Infections and infestations) | 0 | 1 | 1 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 3 | 0
Otitis Externa (Infections and infestations) | 0 | 0 | 1 | 0
Periorbital Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 0 | 0
Sialoadenitis (Infections and infestations) | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 1 | 0
Upper Respiratory Tract InfectionUpper Respiratory Tract Infection (Infections and infestations) | 3 | 1 | 1 | 4
Urinary Tract Infection (Infections and infestations) | 1 | 0 | 3 | 0
Vulvovaginal Candidiasis (Infections and infestations) | 0 | 1 | 0 | 0
Arthropod Bite (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 1
Corneal Abrasion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Epicondylitis (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Facial Bones Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 2 | 1
Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Joint Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Muscle Strain (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 1
Post Procedural Complication (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 1
Post Procedural Discomfort (Injury, poisoning and procedural complications) | 1 | 2 | 1 | 0
Post Procedural Inflammation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Post Procedural Swelling (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 1
Procedural Pain (Injury, poisoning and procedural complications) | 1 | 1 | 2 | 7
Skin Abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Tooth Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 1 | 4 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 2
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Joint Effusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Joint Laxity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Joint Noise (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Joint Range Of Motion Decreased (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Lip Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 2
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0
Lumbar Radiculopathu (Nervous system disorders) | 0 | 0 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0
Renal Failure (Renal and urinary disorders) | 0 | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Menopause (Social circumstances) | 0 | 1 | 0 | 0
Walking Aid User (Social circumstances) | 0 | 0 | 0 | 1
Knee Arthroplasty (Surgical and medical procedures) | 0 | 0 | 1 | 0
Peripheral Vascular Disorder (Vascular disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of Study results will not be made before the first multi-site publication by Sponsor. If no manuscript is submitted within 12 months after the Study's database lock, Investigator may publish Study results if he/she submits all proposed Publications to Sponsor 60 days prior to submission. Investigator shall delete Sponsor's Confidential Information and delay Publication up to 60 days to allow Sponsor to file a patent on Confidential Information in the Publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-17): https://cdn.clinicaltrials.gov/large-docs/44/NCT04129944/Prot_SAP_000.pdf